CLINICAL TRIAL: NCT00916643
Title: Post Marketing Surveillance Study for LDL Apheresis Using H.E.L.P. Therapy
Brief Title: Low-Density Lipoprotein (LDL) Apheresis Using H.E.L.P. Therapy
Acronym: Secura
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B. Braun Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBMI_HELP_Secura
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2014-01

CONDITIONS: Familial Hypercholesterolemia
Keywords: Hypercholesterolemia; FH; LDL-C; CHD
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- H.E.L.P. Secura (Experimental): The H.E.L.P. System is a device composed of multiple modules and their associated disposables which can selectively and continuously remove LDL-cholesterol from plasma by precipitating the LDL-cholesterol with high concentrations of heparin in an acidic buffer and returning the plasma to the patient. Procedure steps:
  1. Flushing the system with normal saline.
  2. Filtering whole blood through a 0.2 micron plasma filter for continuous plasma removal.
  3. Mixing the plasma with an equal volume of acetate buffer containing heparin.
  4. Precipitation of LDL as a complex with heparin.
  5. Removing the LDL-heparin precipitate by continuous circulation through a filter.
  6. Removing heparin with use of a heparin adsorber.
  7. Bicarbonate dialysis and ultrafiltration to produce an LDL-free plasma without excess heparin.
  8. Re-mixing the LDL-free plasma with blood coming from the plasma filter and returning the reconstituted blood to the patient.
  Interventions: Device: HELP Secura (apheresis treatment)

INTERVENTIONS:
Device: HELP Secura (apheresis treatment) — Process is described in Arm (above).

SUMMARY:
The objectives of this post-surveillance study are to continue to evaluate the safety and effectiveness of the H.E.L.P. System. The safety and effectiveness will be assessed by evaluating the occurrence of death, cardiovascular events or interventions, angina, and serious unanticipated adverse effects. Laboratory assessments will be made to document low-density lipoprotein cholesterol (LDL-C) reduction and any effects on other blood components. Quality of life assessments will also be made.

The study will also assess the modifications to the H.E.L.P. System, including:

* use of a single heparin adsorber, instead of two smaller adsorbers;
* change in the supplier of the ultrafilter (from Secon to Toray);
* reduction in the number of blood lines from eleven to nine;
* change from a single-layer to a two-layer precipitate filter.

The safety and efficacy of the device specific to these modifications will be evaluated by comparing the safety and efficacy data from the patient registry to the data from the initial clinical study on the device as originally designed.

DETAILED DESCRIPTION:
H.E.L.P. therapy is indicated for use in treating patients with familial hypercholesterolemia (FH) who have undergone six months of optimal diet and drug therapy and whose LDL-C level remains > 300 mg/dl in the absence of CHD or > 200 mg/dl with documented CHD. These patients are divided into three subgroups of interest:

* Group A: functional hypercholesterolemic homozygotes with LDL-C > 500mg/dl;
* Group B: functional hypercholesterolemic heterozygotes with LDL-C > 300mg/dl;
* Group C: functional hypercholesterolemic heterozygotes with LDL-C > 200mg/dl and documented CHD.

Optimal diet therapy is defined as having received instruction by a trained dietitian in the use of a diet meeting the National Cholesterol Education Program (NCEP) Step 2 criteria (< 30% of calories as fat, < 7% of calories as saturated fat, and < 200 mg of dietary cholesterol per day). Optimal drug therapy is defined as having been tried on at least two separate classes of effective serum LDL-C lowering agents (>15% reduction) as currently available for at least six months. These drugs include hydroxy methyl glutaryl (HMG) CoA reductase inhibitors, fibric acid derivatives, niacin, and anion exchange resins. These agents should be used in combination at maximal doses as tolerated by the patient under the supervision of their treating physician to monitor side effects.

Documented coronary heart disease (CHD) includes documentation of coronary heart disease by coronary angiography or a history of myocardial infarction (MI), coronary artery bypass surgery (CABG), percutaneous transluminal coronary angioplasty (PTCA) or alternative revascularization procedure (e.g., atherectomy or stent), or progressive angina documented by exercise or non-exercise stress test.

The primary criteria for evaluating the safety and effectiveness of the device will be:

* Occurrence of Death

  * cardiovascular deaths
  * non-cardiovascular deaths
* Occurrence of Cardiovascular Events

  * MI - stroke
  * unstable angina - transient ischemic attack (TIA)
  * congestive heart failure - pulmonary embolism
  * arrhythmia - peripheral vascular disease
  * hypertension
* Occurrence of Surgical or Non-Surgical Intervention Procedure of the Treatment of Atherosclerotic Cardiovascular Disease (ASCVD) including:

  * coronary artery bypass graft (CABG) surgery
  * peripheral vascular bypass surgery
  * percutaneous transluminal coronary angioplasty (PTCA)
  * percutaneous transluminal coronary artery bypass graft angioplasty
  * percutaneous transluminal peripheral angioplasty (PTA)
  * coronary atherectomy (device)
  * coronary artery bypass graft atherectomy (device)
  * peripheral atherectomy (device)
  * carotid endarterectomy (non-device)
  * peripheral endarterectomy (non-device)
  * coronary artery laser surgery
  * coronary artery bypass graft laser surgery
  * peripheral vascular laser surgery
  * coronary artery stent placement
  * coronary artery bypass graft stent placement
  * peripheral vascular stent placement
  * repair of atherosclerotic aortic and arterial aneurysms
  * limb amputation for ASCVD
* Frequency and severity of CHD Symptoms:

  * chest pain (angina),
  * shortness of breath
  * claudication
* Use of CHD Medications for treatment of:

  * angina
  * heart failure
  * arrhythmias
  * hypertension
  * hyperlipidemia
* Use of Lipid-Lowering Medications and Other Cardiovascular Medications Concomitantly
* Laboratory Assessments (lipid, lipoprotein, chemistry, and clotting factors)
* Quality of life assessments (SF-36)
* Occurrence of Serious and/or Unanticipated Adverse Events Reported During Treatment (e.g., hypotension, nausea, vomiting, syncope)
* Occurrence of other serious illnesses
* Acute Reduction of LDL-C

ELIGIBILITY:
Inclusion Criteria:

* Adequate venous access
* Laboratory values:

  * Hematocrit 30% or greater
  * platelet count between 100,000 and 1,000,000/ml
* Premenopausal women must be surgically sterilized or be on oral contraceptive therapy and have a negative pregnancy test at the onset of treatment with H.E.L.P.
* Patients have familial hypercholesterolemia and have undergone at least 6 months optimal diet and drug therapy and fit group A, B, or C

Exclusion Criteria:

* Presence of any of the following conditions:

  * untreated hypothyroidism
  * decompensated congestive heart failure
  * major arrhythmia
  * uncontrolled diabetes mellitus
  * any malignancy
  * disorders associated with excessive bleeding (e.g., peptic ulcer and hemophilia)
  * established or suspected intracranial disease which might cause intracranial bleeding if the patient is anticoagulated
  * any other medical disorders which lead the treating physician to believe that H.E.L.P. treatment would not be in the best interest of the patient
  * current treatment with anticoagulants
  * diastolic BP > 100 mmHg recorded in two occasions at least 24 hours apart.
  * patients under 18 years of age
  * positive test for Hepatitis [Type A (IgM) or B] antigen, Hepatitis C antibody, or HIV (or diagnosis of AIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 1999-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 113 patients received over 6,000 combined H.E.L.P. treatments at six sites between 2000-2009.
Groups:
- H.E.L.P. Secura: All patients received the same Treatment Arm for this study. Treatments were conducted up to 3 times per week; treatment sessions typ. 2 hours in length.
  H.E.L.P. is a device composed of multiple modules and associated disposables to selectively and continuously remove LDL-cholesterol from plasma by precipitating the LDL-cholesterol with high concentrations of heparin in an acidic buffer and returning the plasma to the patient.
  1. Flush system with normal saline;
  2. Filter whole blood through 0.2 micron plasma filter for continuous plasma removal;
  3. Mix plasma with equal volume of acetate buffer containing heparin;
  4. Precipitate LDL as a complex with heparin;
  5. Remove LDL-heparin precipitate by continuous circulation through a filter;
  6. Remove heparin with use of a heparin adsorber;
  7. Bicarbonate dialysis and ultrafiltration to produce LDL-free plasma without excess heparin;
  8. Re-mix LDL-free plasma with blood from plasma filter; return reconstituted blood to patient.
Period: Overall Study
Arm/Group | H.E.L.P. Secura
Started | 113
Completed | 113
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | H.E.L.P. Secura
Number analyzed (Participants) | 113
Age, Customized [Number; unit: participants] — Not all sites collected this information.
  participants
    <=18 years | 0
    Between 18 and 65 years | 80
    >=65 years | 13
Sex/Gender, Customized [Number; unit: participants] — Not all site collected this information.
  participants
    Female | 56
    Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 113

OUTCOME MEASURES:

1. Primary Outcome: Occurence of Death
Description: The Categories listed in the table are the Adverse Events (or similar) that resulted in death.
Time Frame: Participants were followed for one (1) year following discontinuation of treatment.
Population: Inclusion was per protocol.
Measure: Number; unit: participants
Arm/Group | H.E.L.P. Secura
Number analyzed (Participants) | 113
participants
  Cancer | 1
  Pneumonia after open heart surgery | 1
  Complications of open-heart surgery | 1
  Coronary artery disease | 1

2. Primary Outcome: Occurrence of Cardiovascular Events and Interventions
Description: Adverse Events reported for Cardiovascular disease not directly related to therapy.
Time Frame: Participants were followed for one (1) year following discontinuation of treatment.
Population: The number of participants for analysis was determined per protocol.
Measure: Number; unit: participants
Arm/Group | H.E.L.P. Secura
Number analyzed (Participants) | 113
participants
  Cardiovascular symptoms during therapy | 16
  Cardiovascular symptoms during therapy (serious) | 9

3. Primary Outcome: Serious Unexpected Adverse Events
Time Frame: Participants were followed for one (1) year following discontinuation of treatment.
Population: The number of participants for analysis was determined per protocol.
Measure: Number; unit: participants
Arm/Group | H.E.L.P. Secura
Number analyzed (Participants) | 113
participants | 0

4. Primary Outcome: Frequency and Severity of CHD Symptoms (Angina)
Description: This is equatable to the incidence of Cardiovascular AEs.
Time Frame: Participants were followed for one (1) year following discontinuation of treatment.
Population: The number of participants for analysis was determined per protocol.
Measure: Number; unit: participants
Arm/Group | H.E.L.P. Secura
Number analyzed (Participants) | 113
participants | 23

ADVERSE EVENTS:
Time Frame: From the end of 1999 through 2009.
Arm/Group | H.E.L.P. Secura
Serious Adverse Events (participants affected / at risk) | 9/113
Other Adverse Events (participants affected / at risk) | 29/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H.E.L.P. Secura (N=113)
Angina Pectoris (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
General Chest Pain (Cardiac disorders) | 5 (5) — Events were reported by patients; but not related to treatment and unsubstantiated through further clinical testing.
Myocardial Infarction (Cardiac disorders) | 1 (1)
Unstable Angina (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H.E.L.P. Secura (N=113)
Chest Pain (Cardiac disorders) | 6 (9)
Clogged Precipitate Filter (General disorders) | 3 (7)
Hypotension (Vascular disorders) | 4 (5)
Poor Blood Flow (Vascular disorders) | 3 (6)
Poor Venous Access (Vascular disorders) | 6 (7)
Venous Infiltration (General disorders) | 4 (4)
Weakness (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Client may use the results of the study for its own teaching,research,education,clinical and publication purposes without the payment of royalties or other fees.Client shall submit to Sponsor for review, a copy of any proposed publication resulting from the Study at least thirty(30)days prior to the estimated date of publication, and if no response is received within thirty(30)days of the date submitted to Sponsor,it will be conclusively presumed that the publication may proceed without delay.